CLINICAL TRIAL: NCT07330232
Title: Periosteal Sutures for Fixation of Composite Bone Graft Substitutes in Guided Bone Regeneration: a Randomized Controlled Clinical Trial
Brief Title: Periosteal Sutures Versus Titanium Tacks for Guided Bone Re-generation in the Aesthetic Zone: a Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Franco Cavalla, Prof. Dr. Franco Cavalla, Associate Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEC-SSA 19/2021
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Dental Implants; Dental Implants , Osseointegration , Marginal Bone Loss , Implant Stability; Maxillary Alveolar Reconstruction
Keywords: Guided bone regeneration; Horizontal ridge augmentation; Anterior maxilla; Aesthetic zone; Dental implant placement; Periosteal sutures
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized controlled clinical trial with a two-arm, parallel-group (parallel assignment) design. Patients requiring horizontal guided bone regeneration (GBR) with simultaneous implant placement in the anterior maxilla were randomized to one of two graft-stabilization approaches: (1) periosteal mattress sutures (S) or (2) titanium tacks (T).
  Both groups received the same core surgical intervention (implant placement in healed ridges + horizontal GBR using a xenogeneic composite collagenated bovine block graft covered with a resorbable collagen membrane, followed by tension-free flap closure). The only between-group difference was the fixation method used to stabilize the graft (titanium tacks vs periosteal mattress sutures).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periosteal mattress sutures for graft/membrane stabilization during GBR with implant placement (Experimental): Guided bone regeneration (GBR) with simultaneous implant placement in the anterior maxilla using a composite xenogeneic collagenated bovine block graft covered by a resorbable collagen membrane. Stabilization is achieved with periosteal mattress sutures to immobilize the graft and membrane, followed by tension-free primary flap closure and standard postoperative care.
  Interventions: Procedure: Periosteal mattress sutures for graft/membrane stabilization in guided bone regeneration Titanium tacks for graft/membrane stabilization in guided bone regeneration
- Titanium tacks for graft/membrane stabilization during GBR with implant placement (Active Comparator): Guided bone regeneration (GBR) with simultaneous implant placement in the anterior maxilla using a composite xenogeneic collagenated bovine block graft covered by a resorbable collagen membrane. Stabilization is achieved with titanium tacks to fix the graft and membrane, followed by tension-free primary flap closure and standard postoperative care.
  Interventions: Procedure: Periosteal mattress sutures for graft/membrane stabilization in guided bone regeneration Titanium tacks for graft/membrane stabilization in guided bone regeneration

INTERVENTIONS:
Procedure: Periosteal mattress sutures for graft/membrane stabilization in guided bone regeneration Titanium tacks for graft/membrane stabilization in guided bone regeneration — Periosteal mattress sutures: Hardware-free stabilization of the graft and collagen membrane using periosteal anchorage sutures to limit micromotion during guided bone regeneration with simultaneous implant placement in the anterior maxilla.
  Titanium tacks: Hardware-based stabilization of the graft and collagen membrane using titanium fixation tacks to achieve rigid immobilization during guided bone regeneration with simultaneous implant placement in the anterior maxilla.

SUMMARY:
This randomized controlled clinical study, titled "Periosteal sutures for fixation of composite bone substitutes in guided bone regeneration: a randomized controlled clinical study," is being conducted at the Dental Unit of Hospital San Camilo and is sponsored/funded by SigmaGraft Biomaterials.

Purpose: The purpose of this study is to evaluate whether using a periosteal stabilization suturing technique improves outcomes in guided bone regeneration in the anterior maxilla when a composite bone graft substitute is used in conjunction with dental implant installation.

What participation involves: Participants will undergo clinical assessments and data collection by the research team according to the study protocol. As part of study-related imaging, participants will receive two cone-beam computed tomography (CBCT) scans, which involve exposure to ionizing radiation. To reduce radiation exposure, CBCT imaging will be performed at a private imaging center rather than using a conventional hospital CT scanner, and participants will use a lead apron for additional protection.

Potential benefits and risks: No direct benefit is expected for participants. However, the information gained may help improve future treatment approaches for patients requiring dental implants in the anterior maxilla with associated bone grafting procedures. The main risks described relate to exposure to ionizing radiation from CBCT imaging, and measures are in place to minimize this exposure.

Privacy and voluntary participation: Participant confidentiality will be protected. Study information will be stored securely with restricted access, and analyses will use de-identified data. Participation is voluntary, and participants may withdraw at any time without penalty or loss of benefits to which they are otherwise entitled.

DETAILED DESCRIPTION:
Guided bone regeneration (GBR) performed simultaneously with dental implant placement is a widely used approach to rebuild deficient alveolar ridges in the anterior maxilla (aesthetic zone). Predictable GBR relies on two key conditions: (1) the creation and maintenance of a stable regenerative compartment that protects the graft during early healing, and (2) tension-free primary soft-tissue closure capable of preserving that compartment throughout the regenerative phase. In clinical practice, graft and membrane stabilization is often achieved using titanium fixation devices (e.g., tacks or pins). While titanium tacks can provide rigid immobilization, they add hardware and procedural steps and may require removal during re-entry procedures. Periosteal mattress sutures have been proposed as a hardware-free alternative for stabilization by anchoring the graft and membrane apically and laterally, potentially limiting micromotion without the need for fixation devices.

This pilot randomized controlled clinical study evaluates whether a periosteal mattress suture technique provides postoperative buccal bone regeneration outcomes comparable to those achieved with titanium tacks when performing horizontal GBR in the anterior maxilla together with implant placement. The study is conducted in a hospital-based periodontics setting and was approved by the appropriate scientific ethics committee. All participants provide written informed consent prior to any study-related procedures, and participation is voluntary.

Study design and setting

This is a parallel-arm, randomized controlled clinical trial conducted at the Periodontics Clinic/Dental Unit of Hospital San Camilo. Eligible patients seeking implant therapy in the anterior maxilla are consecutively screened. Those who require horizontal GBR at the time of implant placement and meet eligibility criteria are invited to participate. Random allocation assigns participants to one of two stabilization approaches used during GBR:

Stabilization with titanium tacks (hardware fixation)

Stabilization with periosteal mattress sutures (hardware-free fixation)

To minimize bias in assessments, clinical data collection and radiographic measurements are performed by trained and calibrated personnel who are not involved in the surgical procedures.

Participants and informed consent Potential participants are adults requiring implant therapy in the anterior maxilla and presenting with horizontal ridge deficiency where simultaneous GBR is clinically indicated. Standard clinical and medical screening is conducted to identify contraindications to implant surgery and/or regenerative procedures. Participation is explained verbally and in writing by a trained investigator, and written informed consent is obtained. Participants may withdraw at any time without penalty or loss of benefits to which they are otherwise entitled.

Interventions and surgical procedures

All implants are placed in healed ridges using a standardized surgical approach. Buccal augmentation is performed using a xenogeneic composite collagenated bovine block graft (deproteinized bovine mineral integrated within a collagen matrix) shaped to the recipient site to restore buccolingual contour. The graft is covered with a resorbable collagen membrane. The two study arms differ only in the method used to stabilize the graft and membrane:

Titanium tack group: The graft and/or membrane is secured using titanium tacks to provide rigid fixation.

Periosteal suture group: Stabilization is achieved using a periosteal mattress suture technique. This approach uses vertically oriented periosteal sutures to immobilize the graft laterally, supplemented by a horizontal mattress suture between flap edges to reduce the risk of apical displacement.

In both groups, flap advancement and closure are performed to achieve tension-free primary closure, using standardized soft-tissue management techniques appropriate for GBR in the aesthetic zone.

Study visits and follow-up After consent, a baseline clinical and radiographic assessment is performed, which includes diagnostic imaging and digital impressions. Participants then undergo implant placement with simultaneous GBR according to the assigned stabilization method. Postoperative follow-up includes early healing assessments and suture management (as clinically indicated), with additional follow-up visits consistent with institutional implant protocols. Long-term healing is evaluated at approximately six months, at which time a follow-up CBCT scan and digital impressions are obtained for quantitative evaluation of regenerated tissues.

Outcomes and assessments (overview) Radiographic outcomes are assessed using standardized cone-beam computed tomography (CBCT) acquisition protocols. Buccal bone dimensions are evaluated around the implant site at predefined reference levels apical to the implant platform, allowing comparison of postoperative buccal bone thickness between groups. A derived measure of the reconstructed buccal bone contour/area across the evaluated region may also be calculated to provide an integrated assessment of the buccal bone envelope. Clinical observations during follow-up (including healing quality and any complications) are documented according to protocol.

Imaging and radiation safety Participation involves two CBCT scans. CBCT imaging uses ionizing radiation; therefore, risk minimization measures are implemented. Imaging is performed using CBCT (rather than a conventional hospital CT scanner) to reduce radiation exposure, and participants use a lead apron to further decrease dose.

Potential benefits and risks Participants are not expected to receive a direct benefit from taking part in the study beyond the standard-of-care implant and GBR procedure they require clinically. The main study-related risk is exposure to ionizing radiation from CBCT imaging; measures are in place to minimize this exposure. Surgical risks are those typically associated with implant placement and guided bone regeneration procedures and are managed according to standard clinical protocols and follow-up.

Confidentiality and data handling Participant confidentiality is maintained throughout the study. Personal identifiers are protected, study records are stored securely with restricted access, and analyses use de-identified data whenever possible. Only authorized study personnel have access to identifiable information, and data are handled according to applicable regulations and institutional policies.

Funding and support The study is funded/supported by the sponsor, who provides the regenerative biomaterials used in the study and covers study-related radiographic examinations and laboratory costs as described in the informed consent documentation.

ELIGIBILITY:
Inclusion criteria

Patients seeking implant therapy in the anterior maxilla.

Patients requiring simultaneous guided bone regeneration (GBR) at the time of implant placement.

Implant placement performed in a healed ridge (not an immediate post-extraction site).

Able and willing to provide written informed consent.

Exclusion criteria

Uncontrolled diabetes.

Ongoing bisphosphonate therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Mean buccal bone thickness (mm) | 6 months
  Buccal bone thickness is measured on CBCT at 1 mm, 3 mm, and 6 mm apical to the implant platform (linear distance from implant surface to the outer buccal bone contour). The primary outcome is the mean of these three measurements for each implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Camilo, San Felipe, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moreno X, Neira P, Mandakovic D, Strauss FJ, Cavalla F. Pilot Study: Periosteal Mattress Sutures as an Alternative to Pins and Screws in Guided Bone Regeneration in the Esthetic Zone. Int J Periodontics Restorative Dent. 2023 Oct 24;(7):s217-s226. doi: 10.11607/prd.6212. PMID 37879059

DOCUMENTS (3):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT07330232/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT07330232/SAP_001.pdf
  • Informed Consent Form (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT07330232/ICF_002.pdf